CLINICAL TRIAL: NCT00446329
Title: Cinacalcet for Secondary Hyperparathyroidism in Patients Receiving Hemodialysis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: due to financial problems
Sponsor: Papageorgiou General Hospital (Other)
Responsible Party: Principal Investigator, Efstathios Mitsopoulos, Nephrologist, Papageorgiou General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 109/16-01-2007
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — Cinacalcet

INTERVENTIONS:
Drug: cinacalcet — Initiation dose of cinacalcet 30 mg/day. Titration every 2-3 weeks with a maximum dose of 180 mg/day.

SUMMARY:
The 1st phase of the study will assess the acute biochemical response of PTH, calcium and phosphorus to orally administered doses of cinacalcet once (60mg) or twice (30mg x 2) per day.

The 2nd phase of the study designed to evaluate the long term effects of cinacalcet on BMD (bone mineral density)and the levels of PTH, calcium, phosphorus as well as its ability to control secondary hyperparathyroidism without simultaneous administration of other vitamin D compounds.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 yrs
* On hemodialysis for at least 3 months (thrice weekly)
* iPTH >300pg/ml or histological evidence of secondary hyperparathyroidism
* Calcium > 8.1 mg/dl

Exclusion Criteria:

* Unstable clinical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-07

PRIMARY OUTCOMES:
Effects of cinacalcet on bone mineral density and bone histology in hemodialysis patients | one year period

CONTACTS AND LOCATIONS:
Overall Officials: Efstathios Mitsopoulos, MD, Principal Investigator — Papageorgiou General Hospital, Thessaloniki, Greece
Locations (1):
- Papageorgiou General Hospital, Thessaloniki, Greece